CLINICAL TRIAL: NCT06768580
Title: Effect of Oral Melatonin Versus Intraoperative Lidocaine Infusion on Incidence of Postoperative Delirium in Elderly Patients Undergoing Total Hip Arthroplasty: Prospective Randomized Controlled Blinded Study
Brief Title: Effect of Oral Melatonin Versus Intraoperative Lidocaine Infusion on Incidence of Postoperative Delirium in Elderly Patients Undergoing Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Alshaimaa Soliman Alasrag, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD277/9/24
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Oral Melatonin; Lidocaine Infusion; Postoperative Delirium; Elderly Patients; Total Hip Arthroplasty
MeSH Terms: conditions — Emergence Delirium | interventions — Melatonin; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Melatonin group (Experimental): Patients will receive one capsule of melatonin (5mg) orally the night before surgery at 9 pm, the night of the operation, and two nights after the surgical operation at 9 pm, also the patients will receive 10 ml bolus of saline intravenous (IV) over 10 min before induction of anesthesia, then continuous infusion of saline (20 ml/hr) until the end of surgery.
  Interventions: Drug: Melatonin
- Lidocaine group (Experimental): Patients will receive a bolus (10 ml) of intravenous lidocaine (1mg/kg) diluted with saline over 10 min before induction of anesthesia. Continuous infusion of 1.5 mg/kg/hr of intravenous lidocaine diluted with saline (20 ml/hr) will be administered until the end of the surgery, also will receive placebo capsule the night before surgery at 9 pm, the night of operation and two nights after the surgical operation at 9 pm.
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): Patients will receive a bolus (10 ml) of saline over 10 min before induction of anesthesia, then continuous infusion of saline (20 ml/hr) and placebo capsule the night before surgery at 9 pm, the night of the operation and two nights after the surgical operation at 9 pm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Patients will receive one capsule of melatonin (5mg) orally the night before surgery at 9 pm, the night of the operation, and two nights after the surgical operation at 9 pm, also the patients will receive 10 ml bolus of saline intravenous (IV) over 10 min before induction of anesthesia, then continuous infusion of saline (20 ml/hr) until the end of surgery.
  Arms: Melatonin group
Drug: Lidocaine — Patients will receive a bolus (10 ml) of intravenous lidocaine (1mg/kg) diluted with saline over 10 min before induction of anesthesia. Continuous infusion of 1.5 mg/kg/hr of intravenous lidocaine diluted with saline (20 ml/hr) will be administered until the end of the surgery, also will receive placebo capsule the night before surgery at 9 pm, the night of operation and two nights after the surgical operation at 9 pm.
  Arms: Lidocaine group
Drug: Placebo — Patients will receive a bolus (10 ml) of saline over 10 min before induction of anesthesia, then continuous infusion of saline (20 ml/hr) and placebo capsule the night before surgery at 9 pm, the night of the operation and two nights after the surgical operation at 9 pm.
  Arms: Control group

SUMMARY:
The aim of this study is to assess the effect of oral melatonin versus intraoperative lidocaine infusion on incidence of postoperative delirium in elderly patients undergoing total hip arthroplasty under spinal anesthesia.

DETAILED DESCRIPTION:
Delirium is defined according to The American Psychiatric Association's fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), as disturbance in attention and awareness developed over a short period of time , its severity tends to fluctuate during the course of a day, these disturbances cannot be better explained by other pre-existing neurocognitive disorders and do not occur in severely reduced arousal level such as coma. Delirium can be further classified into hyperactive, hypoactive and mixed.Postoperative delirium (POD) usually occurs in the recovery room and appears up to 5 days after surgery.

The prevalence of POD in elderly patients undergoing surgery varies from 20% to 45%. Patients undergoing hip fracture surgery are at higher risk of POD than patients undergoing other types of surgery. This may be related to their older age, higher incidence of comorbidities, and greater physical weakness.

Melatonin (N-acetyl-5-methoxytryptamine) is a neurohormone that is discharged by the pineal gland produced from the amino acid tryptophan. Synthetic melatonin has been effectively utilized in the treatment of sleep disorders. It was likewise utilized as a premedication and it provided excellent anxiolysis, sedation, and sympatholytic impacts with the merit of not influencing the patients' cognition in addition to its analgesic effect.

Lidocaine, an amide local anesthetic and class-1 antiarrhythmic with sedative and anti-inflammatory properties, is increasingly used as a part of a multimodal intraoperative anesthetic adjunct in a variety of surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients aged >65 years old undergoing unilateral total hip arthroplasty.
* Patients with body mass index (BMI) (18-30) kg/m2.
* American Society of Anesthesiologists (ASA) physical status I-III, scheduled to undergo unilateral total hip arthroplasty.

Exclusion Criteria:

* History of mental illness or scoring less than 8 using abbreviated mental test (AMT) before operation.
* Obvious sinus bradycardia (heart rate of <50 beats per minute) or other serious cardiovascular diseases.
* Symptomatic cerebrovascular disease (such as previous stroke).
* History of liver and kidney dysfunction.
* Allergy to lidocaine or melatonin.
* Metabolic disorders and fluid, electrolytes disturbances.
* Alcohol dependence or drug abuse.
* Redo surgery or infectious complications.
* CNS medications (antipsychotics, anticonvulsants, antiparkinsonian, antidepressants).
* History of deep vein thrombosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium (POD) | 1st five days postoperatively
  Incidence of postoperative delirium in elderly patients undergoing total hip arthroplasty will be recorded

SECONDARY OUTCOMES:
Severity of delirium | 1st five days postoperatively
  Severity of delirium will be assessed using (CAM-S) score. The sum of the CAM-S scores ranges from 0 to 7 (7 = most severe).
Onset of delirium | 1st five days postoperatively
  The onset of delirium will be recorded.
Duration of delirium | 1st five days postoperatively
  The duration of delirium will be recorded.
Degree of pain | 24 hours postoperatively
  Postoperative pain will be assessed using the visual analogue scale (VAS) score (0 point indicates no pain and 10 indicate maximum pain). Patients will receive epidural analgesia if VAS score is ≥4.
Length of hospital stay | Till the discharge from the hospital (up to 2 weeks).
  Length of hospital stay will be recorded from the admission till the discharge from the hospital.
Adverse effects | 24 hours Postoperatively
  Any undesirable side effects that may occur intraoperatively or postoperatively will be recorded and treated (e.g., nausea, vomiting, bradycardia, hypotension, respiratory depression and local anesthetic toxicity).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author